CLINICAL TRIAL: NCT05875142
Title: Scalable Digital Delivery of Evidence-based Training for Addiction Professionals to Maximize Treatment Admission and Retention Rates of Opioid Use Disorder in Affected Families
Brief Title: Scalable Digital Delivery of Evidence-based Training for Professionals to Maximize Treatment Rates of OUD in Families
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: We The Village, Inc. (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); Public Health Management Corporation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2202; 1R44DA053845-01A1 (NIH)
Record Dates: First submitted 2023-05-16; First posted 2023-05-25 (Actual); Results first posted 2025-01-20 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: Community Reinforcement And Family Training; Family Health; Substance-Related Disorders
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Intervention Model Description: Conduct a pilot study of 3 levels of digital training (Level 1 - Digital tutorial only [T]; Level 2 - Tutorial & digital training materials for self-study [TM]; Level 3 - Tutorial, digital materials, feedback and coaching [TMC]) to establish feasibility, acceptability, and examine the effects of training on CRAFT knowledge, fidelity, and treatment entry and retention.
Who Masked: Outcomes Assessor
Masking Description: The participants will know what group they are in. When data is sent to the statistician for analysis it will be coded in the groups (e.g., 123) without informing which is which. This masks (or blinds) him to the condition.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- T - Digital Tutorial overview (Active Comparator): A digital tutorial consisting of a curriculum dashboard for review of 10(?) modules, including videos, PDFs, text and quizzes, which are to be self-administered over two weeks. Modules remain available during the 10-week post tutorial period. Participants receive weekly contact encouraging engagement in all of the materials available to them.
  Interventions: Behavioral: Behavioral: Digital Tutorial Overview
- TM - Digital Tutorial plus training Materials (Experimental): Participants receive the digital tutorial (T) as described above plus access to 10 modules of digital training materials released weekly over the 10-week post tutorial period.
  Interventions: Behavioral: Behavioral: Digital Tutorial Overview; Behavioral: Behavioral: Training Materials
- TMC - Digital Tutorial plus training Materials plus feedback and Coaching (Experimental): Participants receive the digital tutorial (T) plus the digital Training materials as described in the two arms above plus they submit audio recordings of sessions with clients and receive feedback on their application of CRAFT and coaching on how to improve.
  Interventions: Behavioral: Behavioral: Digital Tutorial Overview; Behavioral: Behavioral: Training Materials; Behavioral: Behavioral: Feedback and Coaching

INTERVENTIONS:
Behavioral: Behavioral: Digital Tutorial Overview — Self study of a digital tutorial covering an overview of CRAFT designed to be reviewed within 2 weeks.
  Other Names: T
Behavioral: Behavioral: Training Materials — 10 weeks post-tutorial access to additional digital training materials.
  Other Names: TM
  Arms: TM - Digital Tutorial plus training Materials; TMC - Digital Tutorial plus training Materials plus feedback and Coaching
Behavioral: Behavioral: Feedback and Coaching — 10 weeks post-tutorial access to additional digital training materials and systematic feedback and coaching.
  Other Names: TMC
  Arms: TMC - Digital Tutorial plus training Materials plus feedback and Coaching

SUMMARY:
The goal of this project is to develop and evaluate the technical feasibility and commercial viability of a scalable digital counselor training program for CRAFT.

This pilot project will develop an enhanced training model for CRAFT and digitize it to maximize scalability. In this project, investigators will:

Aim 1: Produce the digital counselor training prototype and coaching process, tailored to OUD - with stakeholder input.

Aim 2: Conduct a pilot study of 3 levels of digital training (Level 1 - Digital tutorial only [T]; Level 2 - Tutorial & digital training materials for self-study [TM]; Level 3 - Tutorial, digital materials, feedback and coaching [TMC]) to establish feasibility, acceptability, and examine the effects of training on CRAFT knowledge, fidelity, and treatment entry and retention.

DETAILED DESCRIPTION:
The goal of this project is to develop and evaluate the technical feasibility and commercial merit of a scalable digital training program for Community Reinforcement and Family Training (CRAFT). The product would be tailored to prepare counselors to work with family members of treatment-resistant individuals (Identified Persons; IPs) with opioid use disorder (OUD).

We will recruit counselors working in addiction related professions who work with OUD affected populations. We will enroll 15 participants per study arm. Our primary hypothesis addresses feasibility, and our secondary hypotheses involve a Stage 1b pilot study. Therefore, according to Rounsaville and colleagues' "Stage model of behavioral research", the current study is a Stage 1b pilot trial where a sample size of 15-30 per arm is ideal. In the pilot of our CRAFT Family product,15 participants per group was adequate to assess acceptance and feasibility, attain several statistically significant differences between groups and to estimate effect and sample size for a full trial.

We will assign counselors to one of three training groups using a blocked randomization procedure to control for level of education (highschool/GED, bachelors, masters, PhD) and training and experience in CBT and applied behavior analysis (ABA) as CRAFT is a CBT based on ABA principles. We will use an additive components design consisting of: 1) digital tutorial only (T), 2) digital tutorial plus digital training materials (TM), and 3) digital tutorial, digital training materials plus feedback and coaching (TMC). This design will allow us to assess whether the digital training materials improve counselor outcomes relative to the tutorial only, but will not allow us to access their contribution, if any, to the full training product (TMC). We considered adding a group with tutorial, feedback and coaching (TC), but opted for the simpler design. We can determine the contribution of the digital training materials in a future study, if warranted.

The study will be conducted completely digitally, online. Treatment Conditions Digital Tutorial (T) All participants will continue to have access to tutorial materials throughout the study. Participants assigned to the T condition receive ONLY the tutorial. Afterwards they will be encouraged via weekly emails to continue using the resources in the online tutorial to revisit the CRAFT lessons on their own during the 10-week period between post-tutorial and the final assessment.

Digital Tutorial, with training materials (TM) Participants assigned to the TM condition will complete the tutorial and then receive access to the additional training materials. They will not receive any feedback or video-calls for coaching. They will be encouraged via weekly emails to continue to learn CRAFT on their own during the 10-week post-tutorial period by using the new resources in the online tutorial and the digital training materials Digital Tutorial, with training materials plus feedback and coaching (TMC) Systematic feedback and coaching during the 10-week post-tutorial to final assessment period will be provided to only to participants assigned to the TMC condition. Participants will be required to submit audio taped sessions with clients (up to 12 allowed), for which they will digitally receive written feedback and live video-call coaching. Participants will be encouraged to re-submit their audio taped sessions until they meet the criteria needed for certification in the CRAFT procedure or until the phase is over (whichever occurs first).

Participants will receive individual written Personal Performance Feedback on all audio taped sessions that they submit. This feedback is generated by two CRAFT certified coaches (i.e., CRAFT Trainer or CRAFT Coder) who accesses the digitally audio taped sessions via a secure server. The coach listens to the audiotape and records a session content checklist that indicates key procedures for each module. For each key component, the coach indicates whether it was addressed in the session, rates the quality of implementation for that component (1=poor to 5-excellent) and writes comments praising specific behaviors or making suggestions for further improvement. This feedback is password protected and emailed to the counselor. Every week during the intervention period TMC participants will participate in 30-min video-call Coaching Sessions.

All counselors will complete assessments pre-tutorial, post-tutorial, and at 12 weeks post-tutorial. Each assessment point will include a series of questionnaires and a role play with a standardized patient.

Assessing a) acceptability and feasibility (via surveys on training expectations, satisfaction, usefulness and usability, implementation potential, and price sensitivity); and b) knowledge and fidelity (via a knowledge test and direct observation of audiotapes counselor CRAFT sessions).

ELIGIBILITY:
Inclusion Criteria:

* Is over 19
* Lives in the US
* Working in a counselor-related profession
* Has not been trained in CRAFT
* Provides at least 45 minute individual counselor sessions each week to ≥5 clients (CSO or IP)
* If not already providing care to CSOs, is willing and able to do so
* Counseling work involves clients affected by OUDs, or might if they learned CRAFT
* Is able and willing to submit the required session audiotapes and participate in the tutorial and training and intervention activities over the course of the 12-week study
* Reports having access to a computer and smartphone with internet access, email, and word processing capability
* Demonstrates complete understanding of the requirements for participation in the study by reading and signing the consent form
* Provides valid locator information to allow research and CRAFT training staff to contact them to schedule study-related appointments
* Completes the first assessment mock session with our standardized patient (SP) and pre-tutorial surveys

Exclusion Criteria:

* Does not agree to participate
* Does not complete the baseline assessment requirements
* Is not English-speaking
* Participated in the Qualitative Review study

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2023-05-23 (Actual); Primary Completion 2023-09-26 (Actual); Study Completion 2023-09-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jane Macky, MA, Principal Investigator — We The Village, Inc.
Locations (1):
- We The Village, Inc., New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- T - Digital Tutorial Overview: A digital tutorial consisting of a curriculum dashboard for review of 10 modules, including videos, PDFs, text and quizzes, which are to be self-administered over two weeks. Modules remain available during the 10-week post tutorial period. Participants receive weekly contact encouraging engagement in all of the materials available to them.
- TM - Digital Tutorial Plus Training Materials: Participants receive the digital tutorial (T) plus access to 10 modules of digital training materials released weekly over the 10-week post tutorial period.
- TMC - Digital Tutorial Plus Training Materials Plus Feedback and Coaching: Participants receive the digital tutorial (T) plus the digital Training materials (TM) plus they submit audio recordings of sessions with clients and receive feedback on their application of CRAFT and coaching on how to improve.
Period: Overall Study
Arm/Group | T - Digital Tutorial Overview | TM - Digital Tutorial Plus Training Materials | TMC - Digital Tutorial Plus Training Materials Plus Feedback and Coaching
Started | 15 | 16 | 16
Mock Session | 13 | 12 | 12
Completed | 15 | 15 | 15
Not Completed | 0 | 1 | 1
Not completed — Lost to Follow-up | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | T - Digital Tutorial Overview | TM - Digital Tutorial Plus Training Materials | TMC - Digital Tutorial Plus Training Materials Plus Feedback and Coaching | Total
Number analyzed (Participants) | 15 | 16 | 16 | 47
Age, Continuous [Mean (Full Range); unit: years] | 45 [31 to 61] | 45 [28 to 66] | 45 [23 to 70] | 45 [23 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 13 | 8 | 35
  Male | 1 | 3 | 8 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 3 | 1 | 5
  Not Hispanic or Latino | 14 | 12 | 14 | 40
  Unknown or Not Reported | 0 | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 1
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 1
  Black or African American | 1 | 0 | 1 | 2
  White | 12 | 12 | 12 | 36
  More than one race | 2 | 3 | 1 | 6
  Unknown or Not Reported | 0 | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 15 | 16 | 16 | 47
Community Reinforcement And Family Training (CRAFT) Procedure Fidelity [Mean (Full Range); unit: Scores on a scale] — CRAFT performance on the mock sessions was observed by trained coders who rated performance of each CRAFT treatment entry procedure (6 items), homework procedures (2 items), overall CRAFT approach (2 items), and general clinical skill (4 items) on a 5-point scale (i.e., 1 =poor; 3 =satisfactory; 5 =excellent). A total score was calculated by summing across all 14 items for each participant. Average scores were calculated for each participant group at baseline and at 12-week follow-up. Scores could range from 14 - 70 on the overall total. Higher scores indicated better performance.
  Scores on a scale | 33.20 [24 to 42] | 32.50 [28 to 39] | 31.69 [25 to 42] | 32.45 [24 to 42]
Community Reinforcement and Family Training (CRAFT) Knowledge Test [Mean (Full Range); unit: Score on knowledge quiz] — Measuring the proficiency with which participants answer questions about the CRAFT approach.
  The 20-item CRAFT Knowledge Test was scored by calculating the number of correct answers for each individual and then averaging scores across participants within each group (T, TM, TMC). Scores could range from 0 - 20. Higher scores indicate greater knowledge.
  Score on knowledge quiz | 10.3 [5 to 14] | 11.7 [6 to 16] | 9.7 [6 to 15] | 10.57 [5 to 16]
Implementation potential scale (IPS) [Mean (Full Range); unit: Scores on a scale] — Mean Implementation Potential Scores (IPS) scores were computed for each dimension at each assessment point by adding ratings on a 6-point scale (1-6) within each 4 dimensions (Acceptability/Efficacy = 10 items, range 10 - 60; Implementation Commitment = 8 items, range 8 - 48; Administrative Support = 4 items, range 4 - 24; and Organizational Resources = 4 items, range 4 - 24). A single IPS score was calculated by adding all 26 items for overall perceived implementation potential of CRAFT. The total IPS score could range from 26 - 156. Higher scores indicate better implementation potential. Population: Number analyzed is different from overall, as some participants did not complete each item of the IPS measurement and so did not produce an overall IPS score and were not analyzed.
  Scores on a scale
    number analyzed (Participants) | 8 | 9 | 8 | 25
    (all) | 138.1 [97 to 156] | 142.6 [113 to 155] | 136.4 [79 to 156] | 139.0 [79 to 156]

OUTCOME MEASURES:

1. Primary Outcome: Community Reinforcement And Family Training (CRAFT) Procedure Fidelity
Description: CRAFT performance on the mock sessions was observed by trained coders who rated performance of each CRAFT treatment entry procedure (6 items), homework procedures (2 items), overall CRAFT approach (2 items), and general clinical skill (4 items) on a 5-point scale (i.e., 1 =poor; 3 =satisfactory; 5 =excellent). A total score was calculated across all 14 items for each participant. Average scores on each procedure and in total were calculated for each participant group at baseline and at 12-week follow-up. Scores could range from 6 - 30 on treatment entry; 2 - 10 on homework and CRAFT approach; 4 - 20 on general clinical skill; and 14 - 70 on the overall total. Higher scores indicated better performance
Time Frame: 3 months
Measure: Mean (Full Range); unit: Score on a scale
Arm/Group | T - Digital Tutorial Overview | TM - Digital Tutorial Plus Training Materials | TMC - Digital Tutorial Plus Training Materials Plus Feedback and Coaching
Number analyzed (Participants) | 13 | 12 | 12
Score on a scale | 44.00 [34 to 52] | 52.75 [39 to 63] | 57.25 [47 to 66]
Statistical Analysis 1: Comparison: T - Digital Tutorial Overview vs TM - Digital Tutorial Plus Training Materials; T compared with TM; Test type: Non-Inferiority — test of non-inferiority is H0: control>=treatment vs HA: control<treatment; p = 0.0008, t-test, 1 sided
Statistical Analysis 2: Comparison: T - Digital Tutorial Overview vs TMC - Digital Tutorial Plus Training Materials Plus Feedback and Coaching; T compared with TMC; Test type: Non-Inferiority — test of non-inferiority is H0: control>=treatment vs HA: control<treatment; p = 0.00000503, t-test, 1 sided

2. Secondary Outcome: Community Reinforcement and Family Training (CRAFT) Knowledge Test
Description: Measuring the proficiency with which participants answer questions about the CRAFT approach.
  The 20-item CRAFT Knowledge Test was scored by calculating the number of correct answers for each individual and then averaging scores across participants within each group (T, TM, TMC). Scores could range from 0 - 20. Higher scores indicate greater knowledge.
Time Frame: 3 months
Measure: Mean (Full Range); unit: Score on knowledge quiz
Arm/Group | T - Digital Tutorial Overview | TM - Digital Tutorial Plus Training Materials | TMC - Digital Tutorial Plus Training Materials Plus Feedback and Coaching
Number analyzed (Participants) | 14 | 13 | 15
Score on knowledge quiz | 13.0 [5 to 17] | 15.0 [13 to 18] | 15.4 [11 to 18]
Statistical Analysis 1: Comparison: T - Digital Tutorial Overview vs TM - Digital Tutorial Plus Training Materials; T compared with T; Test type: Non-Inferiority — test of non-inferiority is H0: control>=treatment vs HA: control<treatment; p = 0.0176, t-test, 1 sided
Statistical Analysis 2: Comparison: T - Digital Tutorial Overview vs TMC - Digital Tutorial Plus Training Materials Plus Feedback and Coaching; Comparing T with TMC; Test type: Non-Inferiority — test of non-inferiority is H0: control>=treatment vs HA: control<treatment; p = 0.0056, t-test, 1 sided

3. Secondary Outcome: Program Implementation Potential Scale
Description: Measure Description: Mean Implementation Potential Scores (IPS) scores were computed for each dimension at each assessment point by adding ratings on a 6-point scale (1-6) within each 4 dimensions (Acceptability/Efficacy = 10 items, range 10 - 60; Implementation Commitment = 8 items, range 8 - 48; Administrative Support = 4 items, range 4 - 24; and Organizational Resources = 4 items, range 4 - 24). A single IPS score was calculated by adding all 26 items for overall perceived implementation potential of CRAFT. The total IPS score could range from 26 - 156. Higher scores indicate better implementation potential.
Time Frame: 3 months
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | T - Digital Tutorial Overview | TM - Digital Tutorial Plus Training Materials | TMC - Digital Tutorial Plus Training Materials Plus Feedback and Coaching
Number analyzed (Participants) | 10 | 9 | 8
score on a scale | 136 [116 to 154] | 134 [104 to 156] | 134 [86 to 156]
Statistical Analysis 1: Comparison: T - Digital Tutorial Overview vs TM - Digital Tutorial Plus Training Materials; T compared with TM; Test type: Non-Inferiority — test of non-inferiority is H0: control<=treatment vs HA: control>treatment; p = 0.4066, t-test, 1 sided
Statistical Analysis 2: Comparison: T - Digital Tutorial Overview vs TMC - Digital Tutorial Plus Training Materials Plus Feedback and Coaching; T compared with TMC; Test type: Non-Inferiority — test of non-inferiority is H0: control<=treatment vs HA: control>treatment; p = 0.4045, t-test, 1 sided

4. Other Pre Specified Outcome: New Treatment Entry: Identified Patient Treatment Entry Status
Description: Participants report whether their client's loved one has attended any treatment for their opioid use problem since the baseline assessment by answering questions regarding participation in treatment. In addition, reports of treatment entry to WTV staff were categorized as treatment entry. The outcome is the percentage of participants reporting that their client's loved one (identified patient; IP) entered new treatment
Time Frame: 3 months
Measure: Number; unit: Percentage of participants
Arm/Group | T - Digital Tutorial Overview | TM - Digital Tutorial Plus Training Materials | TMC - Digital Tutorial Plus Training Materials Plus Feedback and Coaching
Number analyzed (Participants) | 14 | 14 | 16
Percentage of participants | 23.1 | 48.4 | 80

ADVERSE EVENTS:
Time Frame: Adverse event information was monitored during the intervention, which was 12 weeks for participants from baseline to follow up.
Description: This was a brief, minimal risk study of counselor training methods in a healthy population. Risks were: 1. Breach of confidentiality, 2. Discomfort completing measures, 3. Perceived invasion of privacy, 4. Perceived coercion to participate, 5. Disappointment in random assignment.
  Staff were trained to report AEs and SAEs that were mentioned during digital interactions.
Arm/Group | T - Digital Tutorial Overview | TM - Digital Tutorial Plus Training Materials | TMC - Digital Tutorial Plus Training Materials Plus Feedback and Coaching
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/16 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 0/15 | 0/16 | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2023-03-22): https://cdn.clinicaltrials.gov/large-docs/42/NCT05875142/Prot_000.pdf
  • Statistical Analysis Plan (2023-09-26): https://cdn.clinicaltrials.gov/large-docs/42/NCT05875142/SAP_001.pdf
  • Informed Consent Form (2023-07-22): https://cdn.clinicaltrials.gov/large-docs/42/NCT05875142/ICF_002.pdf